CLINICAL TRIAL: NCT04860076
Title: Open-label, Uncontrolled, Non-Interventional, Retrospective Study to Evaluate Molecular Determinants of Outcome to the Immune Checkpoint Inhibitors (Anti-PD-1/Anti-PD-L1 Monoclonal Antibodies) Treatment for Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asylia Diagnostics BV (Industry)
Responsible Party: Sponsor
Other Study IDs: BR00012020
Record Dates: First submitted 2021-04-23; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Melanoma; Lung Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms | interventions — pembrolizumab; Ipilimumab; Nivolumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pembrolizumab — Standard of care
  Other Names: Ipilimumab; Nivolumab

SUMMARY:
The recent approval of ICB treatments targeting cytotoxic T-lymphocyte antigen 4 (CTLA-4) and programmed cell death-1 (PD-1/PD-L1) by the US Food and Drug Administration has offered an improved treatment chance for a variety of malignant tumors, including those with a particularly poor prognosis. However, a growing number of studies and case reports show that immunotherapy may accelerate tumor progression in a significant subset of patients ranging from 9% to 27% across multiple histologies and lead to so-called hyperprogressive disease (HPD) that leads to a rapid patient death.

During this NIS study, Asylia Diagnostics aims to fill in the first layer of knowledge leading to the identification of predictive biomarkers and biological mechanisms that could be used for the prediction, diagnosis, and treatment of melanoma and NSCLC HPD patients.

The study is a retrospective clinical study. During this study basic historical medical information and scrolls from FFPE-preserved biopsies taken prior to immunotherapy treatment will be collected. The nature of the study is not invasive and non interruptive to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 18-95 y.o.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky >/=70%)
* Histologically or cytologically confirmed melanoma or lung cancer, the grade of the tumor, diagnosed before enrolment into the study.
* Treatment with anti-PD1/anti-PD-L1 drugs and anti-PD1/anti-PD-L1 drugs in combinations with other therapies
* Subjects may have received any number of prior lines of chemotherapy or targeted therapies
* Availability of FFPE tissue samples received prior to any type of antitumor treatment start
* Complete medical records (stage, receptors status, demographic data)

Exclusion Criteria:

* Has had chemotherapy, targeted small molecule therapy, or radiation therapy >30 Gray within 14 days prior to the baseline biopsy or persistent adverse events (AE) related to prior therapy, which have not recovered (i.e., AEs should be ≤Grade 1 or ≤the value collected at baseline) from AEs due to a previously administered intervention
* Any evidence of uncontrolled system pathology, active infections, active bleeding diathesis, renal graft, hepatitis B, C or HIV.
* Autoimmune diseases such as Addison's disease, thyroiditis, lupus (SLE), Sjogren's syndrome, scleroderma, myasthenia gravis, Grave's disease, and Goodpasture's syndrome, requiring active therapy with corticosteroids. If a patient has been taking steroids, at least 2 weeks must have passed since the last dose. Patients with a history of endocrinopathies (e.g. hypothyroidism, adrenal insufficiency, hypopituitarism) are eligible if they are stable on hormone replacement therapy.
* Patients with prior splenectomy, ocular melanoma
* Recent (within 1 year) history of another cancer with the exceptions of non-melanoma skin cancer, superficial bladder cancer, or localized cervical cancer
* Pregnant patients

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects treated by immune checkpoint inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-06-06 (Estimated); Study Completion 2023-06-06 (Estimated)

PRIMARY OUTCOMES:
RECIST | 24 weeks
  Response Evaluation Criteria in Solid Tumours

SECONDARY OUTCOMES:
PFS | 24 weeks
  Progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borcoman E, Kanjanapan Y, Champiat S, Kato S, Servois V, Kurzrock R, Goel S, Bedard P, Le Tourneau C. Novel patterns of response under immunotherapy. Ann Oncol. 2019 Mar 1;30(3):385-396. doi: 10.1093/annonc/mdz003. PMID 30657859
- [Background] Champiat S, Besse B, Marabelle A. Hyperprogression during immunotherapy: do we really want to know? Ann Oncol. 2019 Jul 1;30(7):1028-1031. doi: 10.1093/annonc/mdz184. No abstract available. PMID 31173063
- [Background] Champiat S, Ferrara R, Massard C, Besse B, Marabelle A, Soria JC, Ferte C. Hyperprogressive disease: recognizing a novel pattern to improve patient management. Nat Rev Clin Oncol. 2018 Dec;15(12):748-762. doi: 10.1038/s41571-018-0111-2. PMID 30361681
- [Background] Friedman CF, Proverbs-Singh TA, Postow MA. Treatment of the Immune-Related Adverse Effects of Immune Checkpoint Inhibitors: A Review. JAMA Oncol. 2016 Oct 1;2(10):1346-1353. doi: 10.1001/jamaoncol.2016.1051. PMID 27367787
- [Background] Fuentes-Antras J, Provencio M, Diaz-Rubio E. Hyperprogression as a distinct outcome after immunotherapy. Cancer Treat Rev. 2018 Nov;70:16-21. doi: 10.1016/j.ctrv.2018.07.006. Epub 2018 Jul 18. PMID 30053725